CLINICAL TRIAL: NCT06839820
Title: IRAPID: Infliximab Infusion Rate in Pediatric Inflammatory Bowel Disease. a Randomized Non-inferiority Trial of Infusion Reactions with Infliximab Infusion-rates of 30 Minutes and 60 Minutes
Brief Title: Infliximab Infusion Rates in Pediatric Inflammatory Bowel Disease
Acronym: iRAPID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Charlotte K Knatten, Principal investigator. Consultant, MD, phd at Department of Pediatrics, Akershus University hospital, University Hospital, Akershus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 812756
Record Dates: First submitted 2025-02-10; First posted 2025-02-21 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Infliximab; Infusion; IBD (Inflammatory Bowel Disease); Patient Satisfaction
Keywords: ibd; pediatric ibd; infliximab; infusion rate
MeSH Terms: conditions — Inflammatory Bowel Diseases; Patient Satisfaction; Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: randomized, crossover, non-inferiority open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rapid first (Active Comparator): 4 infusions of infliximab given over 30 minutes, then 4 infusions of infliximab given over 60 minutes. Totally 8 infusions of infliximab is given during the study, according to the randomized cross-over design.
  Interventions: Other: Infusion rate of infliximab
- Slow infusion first (Active Comparator): 4 infusions of infliximab given over 60 minutes, then 4 infusions of infliximab given over 30 minutes.
  Totally 8 infusions of infliximab is given during the study, according to the randomized cross-over design.
  Interventions: Other: Infusion rate of infliximab

INTERVENTIONS:
Other: Infusion rate of infliximab — Infusion reactions of infliximab is compared between 30 and 60 minutes infliximab infusion-rates.

SUMMARY:
OBJECTIVES OF THE STUDY

1. Investigate whether there are just as few infusion reactions with infliximab infusions of 60 min and 30 min.
2. Investigate patient and nurse satisfaction with infusions of 60 min and 30 min.
3. Investigate resource use in terms of total length of stay and use of nursing resources.

DETAILED DESCRIPTION:
Our primary objective in this study is to compare the incidence of infusion reactions of Infliximab when administered over 30 minutes versus 60 minutes. We hypothesize that there will be no significant differences between the two groups, demonstrating that 30-minute infusions are as safe and effective as the current standard of 60-minute infusions.

Secondary endpoints include evaluating patient and nurse satisfaction with both infusion rates, as well as assessing resource utilization by measuring total outpatient clinic stay and nursing staff allocation.

Additionally, we will explore whether satisfaction, infusion reactions and treatment effectiveness (asessed through clinical scoring systems, endoscopic findings and laboratory results) are affected by patient demographics (such as age, sex), disease type, infusion frequency, or co-treatment with immunomodulators.

Project methodology Study design and implementation Strategy The iRAPID study is designed as a prospective, randomized, open-label, non-inferiority crossover trial designed to compare the safety and effectiveness of 30-minute versus 60-minute infliximab infusions in pediatric IBD patients. The study will be conducted at the Akershus University Hospital Pediatric and Adolescent Outpatient Clinic, where all included patients already receive infliximab infusions for inflammatory bowel disease (IBD). Patients included in the study will be randomized to receiving four consecutive fast 30-minute infusions, or four consecutive standard 60-minute infusions, after which they will switch to the alternative regimen. Each patient will serve as their own control. Randomization will be performed using a validated computer-generated randomization program.

If the patient meets inclusion and exclusion criteria, they will be invited to participate in the study. Written consent will be obtained from parents for children under the age of 16, while patients aged 16 years or older will provide their own written consent. Participation is voluntary, and one may withdraw from the study and return to the standard infusion rate of 60 minutes at any time. Based on the power calculation, 60 patients will be included in the study. This sample size allows for adjustments in dosing, intervals, and concomitant medication according to standard clinical criteria, as well as a safety margin for dropouts.

Infusion reactions will be monitored by an experienced IBD-nurse before, during and after each infusion. Infusion reactions will be dichotomized as yes or no, and categorized as mild/localized, moderate or severe using predefined clinical criteria (See references Lichtenstein, J Crohns Colitis. 2015;9(9):806-15 and Jagt et al, J Pediatr Gastroenterol Nutr. 2023;77(3):373-80). The criteria are based on age-appropriate values from the Pediatric Early Warning Score (PEVS), which ensures consistency in event classification and facilitates reliable safety assessments. The nurse will record vital signs, including pulse, blood pressure and respiratory rate, in addition to observe for symptoms of an infusion reaction, in accordance with the already established standard procedure for infliximab infusions.

* Criteria for mild/localized infusion reaction: Transient and short-lived pruritus, flushing (facial erythema), myalgia or low-grade fever (37.5-37.9°C).
* Criteria for moderate infusion reaction: Fever (temperature >38°C), tachycardia (increase in heart rate >20 beats/min above age-appropriate values in the PEVS chart), sensation of breathlessness or chest tightness or angioedema.
* Criteria for severe infusion reaction: Bronchospasm or laryngospasm, decreased consciousness, hypotension (a drop in systolic blood pressure >20 mmHg from the normal value in the PEVS chart) or anaphylactic shock.

If an infusion reaction occurs, the patient will be assessed with a doctor, and appropriate intervention will follow standard clinical guidelines (Ref Lichtenstein, J Crohns Colitis. 2015;9(9):806-15). In case of an infusion reaction, clinical judgment will be used to assess whether there is an identifiable cause, whether the patient should continue the medication, whether additional treatment is necessary, and how the next infusion should be conducted. All adverse events, including symptoms, interventions, and assessments will be documented in the medical record and the study database.

* In the case of a mild infusion reaction, the infusion rate will be reduced and then gradually increased if tolerated.
* In the case of a moderate infusion reaction, the infusion will be stopped, pharmacological interventions will be considered and if the patient is deemed stable, the infusion will restart at a slower rate with gradual escalation.
* In the case of a severe infusion reaction, the infusion will be stopped immediately, and appropriate treatment will be administered.

Demographic data are recorded to describe the enrolled patients, including age, sex, weight and height, and disease-specific information such as IBD type, duration and extent, and previous treatment including other immunosuppressive treatment, treatment efficacy, and the duration and number of doses of infliximab therapy prior to study inclusion. At each infusion visit, the doctor will also document infliximab dose, infusion interval, and drug concentration. As part of the routine consultation, disease activity will be assessed using validated scoring systems: PUCAI for ulcerative colitis and short-PCDAI for Crohn's disease. Adjustments to treatment intervals and dosing will be made based on clinical jugdements and patient needs, independent of study participation.

Satisfaction will be evaluated using a custom-designed questionnaire completed by patients, parents and nurses. This assessment will provide qualitative insights into the impact of infusion time on both patient/caregiver experience and the clinical workflow.

The economic impact of infusion-rate will be assessed by recording:

* Total time spent in the outpatient clinic from arrival to discharge
* Total nursing time required for each infusion, including preparatory tasks (blood sampling, IV placement), infusion administration, monitoring of the patient and documentation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric IBD patients on infliximab
* 1-17 years
* Received at least 5 infusions of infliximab prior to entry in the study

Exclusion Criteria:

* Receiving infliximab for non-IBD condition (reumatological or other causes)
* previous severe infliximab infusion reaction
* need for an interpreter
* heart failure with hemodynamic impact
* unwillingness to participate

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of infusion reactions with infliximab infusions given over 60 minutes compared to 30 minutes. | depending on patients infusion intervals; 4 weeks x8 = 32 weeks, 8 weeks interval x8 = 64 weeks. The estimated time frame to complete the study for all included patients is april 2026.
  A randomized non-inferiotity trial designed to investigate whether there are just as few infusion reactions with infliximab-infusions given over standard 60 minutes as with 30 minutes infusion rate. All patients receive 8 infliximab infusions during the study. They are randomized either to a) 4 infliximab infusions over 30 minutes first and then 4 inflimab infusions over 60 minutes, or B) 4 infliximab infusions over 60 minutes first and then 4 inflimab infusions over 30 minutes. Each patients receive an infusion interval between 4 to 8 weeks, that is tailered to their disease and needs as judged by the clinician. Data will be collected through study completion (8 infusions), with a time frame between a total of 32 weeks til 64 weeks, depending on the patients infliximab infusion intervals. All infusions reactions that occur during the time frame of these 8 infusions will be included in the analysis.

SECONDARY OUTCOMES:
Investigate patient satisfaction with infliximab infusions of 60 minutes and 30 minutes | During the 8 infliximab infusions, with a time frame between 32 weeks til 64 weeks, depending on the patients infliximab infusion intervalls that may range from every 4th to every 8th week.
  Patient and parental satisfaction with infusion rate is measured on a 10point scale, one question for patients and one for the parents. Patients og parents will be asked every time during the 8 infusions, and all data will be summarized to be included in the analysis a median score for 30 minutes infusions, and 60 minutes infusion. The score will be compared between 30 minutes infusions and 60 minutes infusions to see if there is any difference in satisfaction.
Investigate nurse satisfaction with infliximab infusions of 60 minutes and 30 minutes | During the 8 infliximab infusions, with a time frame between 32 weeks til 64 weeks, depending on the patients infliximab infusion intervalls that may range from every 4th to every 8th week.
  Nurses satisfaction with infusion rate is measured on a 10point scale,. Nurses are asked to rate their satisfaction every time during the 8 infusions, and all data will be summarized to be included in the analysis a median score for 30 minutes infusions, and 60 minutes infusion. The score will be compared between 30 minutes infusions and 60 minutes infusions to see if there is any difference in satisfaction. The overall score of nurse satisfaction will be assessed against factors that may influence the nurses satisfaction, including perceived workload for 30 and 60 minutes infusions (0 -10 score) and if the infusion rate affected chair capasity (0 (very negatively) -10 (very positive) score).
Investigate resource use in terms of total length of stay and costs | During the 8 infliximab infusions, with a time frame between 32 weeks til 64 weeks, depending on the patients infliximab infusion intervalls that may range from every 4th to every 8th week.
  Patients are asked to fill in the time when they arrived and when they left hospital, to assess time spent in hospital for each infusion. Nurses fill out a form to assess time spent for practical administration of medication to the patient. Nurses and patients will be asked every time during the 8 infusions, and all data will be included in an analysis of costs with 30 and 60 minutes infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Akershus University Hospital REK comittee, Study Chair — Akerhus University Hospital
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No
Not allowed due to norwegian goverment

REFERENCES:
- [Background] Lichtenstein L, Ron Y, Kivity S, Ben-Horin S, Israeli E, Fraser GM, Dotan I, Chowers Y, Confino-Cohen R, Weiss B. Infliximab-Related Infusion Reactions: Systematic Review. J Crohns Colitis. 2015 Sep;9(9):806-15. doi: 10.1093/ecco-jcc/jjv096. Epub 2015 Jun 19. PMID 26092578
- [Background] Jagt JZ, Galestin SE, Claesen J, Benninga MA, de Boer NKH, de Meij TGJ. Safety of Accelerated Infliximab Infusions in Children With Inflammatory Bowel Disease: A Retrospective Cohort Study. J Pediatr Gastroenterol Nutr. 2023 Sep 1;77(3):373-380. doi: 10.1097/MPG.0000000000003865. Epub 2023 Jun 15. PMID 37319101
- [Background] Fukuyo S, Saito K, Yamaoka K, Sawamukai N, Hirata S, Nawata M, Iwata S, Tanaka Y. Efficacy and safety of reducing duration of infliximab infusion. Mod Rheumatol. 2014 Mar;24(2):275-80. doi: 10.3109/14397595.2013.843747. Epub 2013 Oct 11. PMID 24251990
- [Background] Neef HC, Riebschleger MP, Adler J. Meta-analysis: rapid infliximab infusions are safe. Aliment Pharmacol Ther. 2013 Aug;38(4):365-76. doi: 10.1111/apt.12389. Epub 2013 Jul 1. PMID 23815183
- [Background] El-Matary W, Dykes DMH, Bauman L, Elkadri A, Carroll MW, Izaguirre MR, deBruyn J, Samson CM, Crim AM, Ali S, Grossman A. Rapid Infliximab Infusion in Children with Inflammatory Bowel Disease: A Multicenter North American Experience. Inflamm Bowel Dis. 2017 Dec;23(12):2104-2108. doi: 10.1097/MIB.0000000000001259. PMID 29140940
- [Background] Bohra A, Rizvi QA, Keung CYY, Vasudevan A, van Langenberg DR. Transitioning patients with inflammatory bowel disease from hospital-based to rapid home-based infliximab: A stepwise, safety and patient-orientated process towards sustainability. World J Gastroenterol. 2020 Sep 28;26(36):5437-5449. doi: 10.3748/wjg.v26.i36.5437. PMID 33024395